CLINICAL TRIAL: NCT04291599
Title: Initial Pain Management in Pediatric Pancreatitis: Opioid vs. Non-Opioid
Acronym: PATIENCE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate patients recruited. Completion of funding
Sponsor: Boston Children's Hospital (Other)
Collaborators: The National Pancreas Foundation (Other)
Responsible Party: Principal Investigator, Amit Grover, Principal Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P00034168
Record Dates: First submitted 2020-02-03; First posted 2020-03-02 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Acute Pancreatitis
Keywords: Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Ketorolac; Ketorolac Tromethamine; Analgesics, Opioid; Morphine; Hydromorphone

STUDY DESIGN:
Intervention Model Description: This will be a phase 2, single-center, unblinded randomized controlled pilot trial of two arms comparing opioid-sparing analgesia to the current BCH institutional practice which has been reported to predominantly include administration of opioids as a first-line analgesic to pediatric patients who present to the emergency department with a diagnosis of acute pancreatitis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental Arm - Ketorolac (Opioid-Sparing) (Experimental): Patients assigned to this arm of the study will follow the standardized step-up approach to pain management per the hospital Evidenced Based Guideline (EBG). If analgesia is not obtained with first-line medications such as acetaminophen, the patient will be given the NSAID ketorolac intravenously every 6 hours at the standard weight-based dose throughout hospitalization. If the patient experiences continued pain, they (or their guardian/ caregiver) may request a rescue medication in the form of low-dose morphine (or an alternative opioid if allergic to morphine) at 0.025 mg/kg/dose every 4 hours.
  Interventions: Drug: Ketorolac
- Control Arm - Conventional Treatment/Standard of Hospital Care (Active Comparator): Patients assigned to this arm of the study will be treated per institutional policy and procedural care as dictated by established hospital order sets and at the discretion of the provider. This may involve the step-up approach per the hospital EBG utilizing acetaminophen or ibuprofen as first-line agents; however, it remains at the discretion of the treating provider. The current standard of care for children presenting to the ED is based on prescribing order sets within the electronic medical record (EMR). Physicians in the BCH emergency department choose in an intermittently-prescribed manner, standard doses of analgesia including acetaminophen (Tylenol) or ibuprofen per the hospital EBG, as well as opioids (morphine, hydromorphone).
  Interventions: Drug: Opioid

INTERVENTIONS:
Drug: Ketorolac — Subjects will be randomized to either receive opioid (standard of care) or opioid-sparing analgesia.
  Other Names: Toradol
  Arms: Experimental Arm - Ketorolac (Opioid-Sparing)
Drug: Opioid — Subjects will be randomized to either receive opioid (standard of care) or opioid-sparing analgesia
  Other Names: Morphine, hydromorphone
  Arms: Control Arm - Conventional Treatment/Standard of Hospital Care

SUMMARY:
This will be a phase 2, single-center, unblinded randomized controlled pilot trial of two arms comparing opioid-sparing analgesia to the current Boston Children's Hospital institutional practice which has been reported to predominantly include administration of opioids as a first-line analgesic to pediatric patients who present to the emergency department with a diagnosis of acute pancreatitis (AP). This is a pilot trial for which many outcomes have not previously been studied in the pediatric AP population. The focus of this investigation will be to investigate the magnitude and variability of effect sizes for designing a future multi-center, double-blinded randomized controlled trial.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is the most common pancreatic disease of childhood with an increasing incidence estimated at 13.2 cases in 100,000 children per year. Given the dearth of pediatric literature, most pediatric providers often rely on diagnostic, prognostic and treatment guidelines that have been derived from adults. This is problematic because adult therapeutic guidelines fail to consider the unique age-related responses and requirements of childhood. Pain management is one of the cornerstones in the treatment of pancreatitis, with abdominal pain being the most common presenting symptom of AP. Currently, there are no data on optimal pain management in pediatric AP. Older guidelines suggest that the "use of intravenous patient-controlled analgesia (PCA) is advantageous" as it allows the patient to self-administer opioids and strike a balance between analgesia and side effects. This requires cognitive maturity to understand how to use PCA and poses challenges for younger children, particularly infants and toddlers, as well as pediatric patients with developmental delay. It is particularly concerning that greater than 94% of surveyed pediatric practitioners would use morphine or related opioids as a first-line therapy in children with AP especially when there have been no studies examining the benefits/risks of opioid vs non-opioid analgesics or opioid-sparing therapies in pediatric AP. Furthermore, we recently reported a retrospective analysis demonstrating that opioids are prescribed far more frequently either alone or in combination with non-opioids (70%) than non-opioid alternatives alone (30%). Amongst all types of analgesia prescribed to children who presented to the BCH emergency department (ED) with acute pancreatitis, morphine was the most common. Further research in this area is imperative, particularly given the recent opioid epidemic. From a pediatric perspective, it has been demonstrated that adolescents are amongst those at risk for opioid abuse, thus there is an urgent need to determine whether opioids are necessary for the management of pain in this vulnerable population with AP.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who present to the ED and are admitted to BCH with a diagnosis of acute pancreatitis or an acute bout of chronic pancreatitis based on INSPPIRE14 Criteria (Appendix 1)
2. Age ≤21 years
3. Patient weight ≥8 kg

Exclusion Criteria:

1. Allergy to morphine (and hydromorphone) or aspirin/NSAID
2. History of renal or hepatic insufficiency
3. History of peptic ulceration
4. History of bleeding diathesis
5. Pregnant females
6. Patients who have a documented history of substance abuse disorder or those who use opioids chronically
7. Patients admitted to the Intensive Care Unit (ICU)
8. Patients who received intravenous opioid patient-controlled analgesia (PCA) in transit or during their ED admission.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Efficacy: amount of opioid analgesia (mg/kg/hr) from the time of enrollment until discharge home, transfer to the ICU, or initiation of PCA | time of enrollment through study completion (approximately 5 days), or transfer to the ICU or initiation of PCA
  The primary endpoint for efficacy is the amount of opioid analgesia (mg/kg/hr) from the time of enrollment until discharge home, transfer to the ICU, or initiation of PCA.

SECONDARY OUTCOMES:
Safety: number of hours from the time of enrollment until discharge home, transfer to the ICU, or initiation of PCA | time of enrollment through study completion (approximately 5 days), or transfer to the ICU or initiation of PCA
  The secondary endpoint for safety is defined as the total number of incident adverse events, grade 2 or higher, from the time of enrollment until discharge home, transfer to the ICU, or initiation of PCA.
Length of stay | time of enrollment through study completion (approximately 5 days), or transfer to the ICU or initiation of PCA
  The secondary endpoint for length of stay is defined as the number of hours from the time of enrollment until discharge home, transfer to the ICU, or initiation of PCA.
Time to initiation of oral or enteral diet | time of enrollment through study completion (approximately 5 days), or transfer to the ICU or initiation of PCA
  The secondary endpoint for time to initiation of oral or enteral diet is defined as the number of hours from the time of enrollment until first oral or enteral intake. The number of hours will be expressed to two decimal places to account for fractions of an hour.
Predefined Feasibility Outcomes to Assess Trial Success | duration of trial, approximately 1 year from the start of enrollment
  The secondary endpoint for feasibility is defined as (1) ≥80% of eligible patients approached for consent during the trial, and (2) ≥20% of eligible patients randomized into the trial.
Pain resolution: pain scores | time of enrollment through study completion (approximately 5 days), or transfer to the ICU or initiation of PCA
  To compare pain resolution from time of enrollment throughout hospital stay by comparing pain scores in patients receiving opioid-sparing therapies to those receiving standard of care opioid analgesics.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Grover, MB BCh BAO, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banks PA, Freeman ML; Practice Parameters Committee of the American College of Gastroenterology. Practice guidelines in acute pancreatitis. Am J Gastroenterol. 2006 Oct;101(10):2379-400. doi: 10.1111/j.1572-0241.2006.00856.x. No abstract available. PMID 17032204
- [Background] Grover AS, Mitchell PD, Manzi SF, Fox VL. Initial Pain Management in Pediatric Acute Pancreatitis: Opioid Versus Non-opioid. J Pediatr Gastroenterol Nutr. 2018 Feb;66(2):295-298. doi: 10.1097/MPG.0000000000001809. PMID 29077648
- [Background] Wu BU, Banks PA. Clinical management of patients with acute pancreatitis. Gastroenterology. 2013 Jun;144(6):1272-81. doi: 10.1053/j.gastro.2013.01.075. PMID 23622137
- [Background] Forsmark CE, Baillie J; AGA Institute Clinical Practice and Economics Committee; AGA Institute Governing Board. AGA Institute technical review on acute pancreatitis. Gastroenterology. 2007 May;132(5):2022-44. doi: 10.1053/j.gastro.2007.03.065. No abstract available. PMID 17484894
- [Background] Rudd RA, Seth P, David F, Scholl L. Increases in Drug and Opioid-Involved Overdose Deaths - United States, 2010-2015. MMWR Morb Mortal Wkly Rep. 2016 Dec 30;65(50-51):1445-1452. doi: 10.15585/mmwr.mm655051e1. PMID 28033313
- [Background] Munro HM, Walton SR, Malviya S, Merkel S, Voepel-Lewis T, Loder RT, Farley FA. Low-dose ketorolac improves analgesia and reduces morphine requirements following posterior spinal fusion in adolescents. Can J Anaesth. 2002 May;49(5):461-6. doi: 10.1007/BF03017921. PMID 11983659
- [Background] Howard ML, Isaacs AN, Nisly SA. Continuous Infusion Nonsteroidal Anti-Inflammatory Drugs for Perioperative Pain Management. J Pharm Pract. 2018 Feb;31(1):66-81. doi: 10.1177/0897190016665539. Epub 2016 Aug 31. PMID 27580638
- [Background] Hadland SE, Wood E, Levy S. How the paediatric workforce can address the opioid crisis. Lancet. 2016 Sep 24;388(10051):1260-1. doi: 10.1016/S0140-6736(16)31573-2. No abstract available. PMID 27673455
- [Background] Bai HX, Lowe ME, Husain SZ. What have we learned about acute pancreatitis in children? J Pediatr Gastroenterol Nutr. 2011 Mar;52(3):262-70. doi: 10.1097/MPG.0b013e3182061d75. PMID 21336157
- [Background] Nydegger A, Heine RG, Ranuh R, Gegati-Levy R, Crameri J, Oliver MR. Changing incidence of acute pancreatitis: 10-year experience at the Royal Children's Hospital, Melbourne. J Gastroenterol Hepatol. 2007 Aug;22(8):1313-6. doi: 10.1111/j.1440-1746.2007.04936.x. Epub 2007 Apr 19. PMID 17489962
- [Background] Morinville VD, Barmada MM, Lowe ME. Increasing incidence of acute pancreatitis at an American pediatric tertiary care center: is greater awareness among physicians responsible? Pancreas. 2010 Jan;39(1):5-8. doi: 10.1097/MPA.0b013e3181baac47. PMID 19752770
- [Background] Abu-El-Haija M, Lin TK, Palermo J. Update to the management of pediatric acute pancreatitis: highlighting areas in need of research. J Pediatr Gastroenterol Nutr. 2014 Jun;58(6):689-93. doi: 10.1097/MPG.0000000000000360. PMID 24614126
- [Background] Miech R, Johnston L, O'Malley PM, Keyes KM, Heard K. Prescription Opioids in Adolescence and Future Opioid Misuse. Pediatrics. 2015 Nov;136(5):e1169-77. doi: 10.1542/peds.2015-1364. PMID 26504126
- [Background] Morinville VD, Husain SZ, Bai H, Barth B, Alhosh R, Durie PR, Freedman SD, Himes R, Lowe ME, Pohl J, Werlin S, Wilschanski M, Uc A; INSPPIRE Group. Definitions of pediatric pancreatitis and survey of present clinical practices. J Pediatr Gastroenterol Nutr. 2012 Sep;55(3):261-5. doi: 10.1097/MPG.0b013e31824f1516. PMID 22357117
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Cohen J. A power primer. Psychol Bull. 1992 Jul;112(1):155-9. doi: 10.1037//0033-2909.112.1.155. PMID 19565683
- [Background] Huguet A, Stinson JN, McGrath PJ. Measurement of self-reported pain intensity in children and adolescents. J Psychosom Res. 2010 Apr;68(4):329-36. doi: 10.1016/j.jpsychores.2009.06.003. Epub 2009 Oct 2. PMID 20307699